CLINICAL TRIAL: NCT05595902
Title: Determination of Normative Values of Navicular Height and Navicular Drop Amount in Geriatric Individuals and Investigation of the Effect of Age, Gender and Body Mass Index on Normative Values
Brief Title: Normative Value for Navicular Drop Test in Older Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Nilufer Kablan, PhD., Asisst. Prof., Istanbul Medeniyet University
Other Study IDs: IstanbulMU81
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Young older adults: ≥65-<75 years of age
- Older adults: ≥75-<90 years of age
- ≥90 years old

SUMMARY:
The aim of this study is to determine the normative values of navicular height and navicular drop in individuals over 65 years of age. The secondary aim is to investigate the effects of age, gender, and body mass index on these normative values.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older
* Having a body mass index between 18.5 and 29.0 kg/m2

Exclusion Criteria:

* Having chronic diseases that affect the foot structure and connective tissue (such as diabetes mellitus, rheumatoid arthritis, gout, etc.).
* Have had foot or ankle surgery in the last 6 months
* Having orthopedic or neurological deformities (related to stroke, Parkinson's, multiple sclerosis, spinal cord injury, etc.) that will affect the foot structure and mobility.
* Dependence on standing and ambulation (except independence gained through the use of assistive devices)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy older adults
Sampling Method: Non-Probability Sample
Enrollment: 445 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
Navicular Drop Test | 10 minutes
  The navicular height and the amount of navicular drop will be made separately for each foot. The navicular prominence is found by palpation and marked with a marker pen when the individual is in a sitting position with the hips and knees flexed to 90 degrees and the subtalar joint in neutral position (the subtalar joint is palpated and the talus is in a neutral position). The height of the navicular protrusion from the ground is measured with a rigid ruler. Then, while the person stands on both feet equally, the height of the navicular protrusion from the ground is also measured with a ruler. The difference between the two measurements is noted as the amount of "navicular drop" (NDT).

SECONDARY OUTCOMES:
Age | 1 minute
  Age
Gender | 1 minute
  Gender
Body-Mass index | 3 minutes
  weight/ (height)2
Foot Posture Index | 15 minutes
  FPI

IPD SHARING:
Plan to Share IPD: No